CLINICAL TRIAL: NCT05794776
Title: Effect of BurstDR and Tonic Spinal Cord Stimulation (SCS) on Glucose Metabolism in Patients With Neuropathic Pain
Brief Title: Effect of Spinal Cord Stimulation (SCS) on Insulin Secretion in Humans
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled anymore
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 047/2022BO2
Record Dates: First submitted 2023-02-17; First posted 2023-04-03 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2023-02

CONDITIONS: Spinal Cord Stimulation; Insulin Secretion

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BurstDR stimulation (Experimental): BurstDR spinal cord stimulation during hyperglycemic clamp
  Interventions: Device: BurstDR stimulation
- Tonic stimulation (Experimental): Tonic spinal cord stimulation during hyperglycemic clamp
  Interventions: Device: Tonic stimulation
- No stimulation (Placebo Comparator): No spinal cord stimulation during hyperglycemic clamp
  Interventions: Device: No stimulation

INTERVENTIONS:
Device: BurstDR stimulation — BurstDR spinal cord stimulation
  Arms: BurstDR stimulation
Device: Tonic stimulation — Tonic spinal cord stimulation
  Arms: Tonic stimulation
Device: No stimulation — Stimulator is switched off
  Other Names: No spinal cord stimulation
  Arms: No stimulation

SUMMARY:
This trial investigates the effect of BurstDR and tonic spinal cord stimulation (SCS) on glucose metabolism and heart rate variability in patients with neuropathic pain.

DETAILED DESCRIPTION:
This study investigates the effect of spinal cord stimulation (BurstDR stimulation versus tonic stimulation versus no stimulation) on glucose metabolism, insulin secretion and heart rate variability in patients with neuropathic pain. To assess insulin secretion, hyperglycaemic clamps are performed in 10 patients. Three different stimulation conditions (BurstDR, tonic and no stimulation) are tested in 10 hyperglycaemic clamps each. A total of 30 clamps are carried out.

ELIGIBILITY:
Inclusion Criteria:

* implanted BurstDR spinal cord stimulating system
* body mass index 18-25 kg/m2

Exclusion Criteria:

* neurological and psychatric diseases
* decompensated diabetes mellitus
* hemoglobin < 13 g/dl
* thrombocytopenia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03-16 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
First and second phase of insulin secretion | Insulinsecretion during clamp (2 hours)
  Modulation of insulin secretion by spinal cord stimulation

SECONDARY OUTCOMES:
Root Mean Square of Successive Differences (RMSSD) | Heart rate variablity during stimulation (10 minutes)
  Modulation of heart rate variability by spinal cord stimulation assessed by electrocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Morgalla, Prof., Principal Investigator — Universitaetsklinikum Tuebingen
Locations (1):
- University Hospital Tuebingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No